CLINICAL TRIAL: NCT00378560
Title: V501 Phase II Efficacy Study in Women Aged 18 to 26
Brief Title: V501 Efficacy Study in Women Aged 18 to 26 (V501-027)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V501-027; 2006_032
Record Dates: First submitted 2006-09-18; First posted 2006-09-20 (Estimated); Results first posted 2010-06-29 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: HPV Infections
MeSH Terms: conditions — Papillomavirus Infections | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Placebo Comparator): Placebo
  Interventions: Biological: Comparator: Placebo
- 2 (Experimental): Vaccine
  Interventions: Biological: Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine

INTERVENTIONS:
Biological: Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine — V501; Gardasil, 0.5 ml injection in 3 dosing regimen
  Other Names: V501; Gardasil
  Arms: 2
Biological: Comparator: Placebo — Placebo 0.5 ml injection in 3 dosing regimen
  Arms: 1

SUMMARY:
A study to evaluate the efficacy, immunogenicity, safety and tolerability of V501 in adult women

ELIGIBILITY:
Inclusion Criteria:

* Female Subject Aged 18 To 26 Years
* With 1-4 Lifetime Sexual Partners

Exclusion Criteria:

* Male Subject

Ages: 18 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1021 (Actual)
Dates: Start 2006-06-12 (Actual); Primary Completion 2009-09-16 (Actual); Study Completion 2009-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Yoshikawa H, Ebihara K, Tanaka Y, Noda K. Efficacy of quadrivalent human papillomavirus (types 6, 11, 16 and 18) vaccine (GARDASIL) in Japanese women aged 18-26 years. Cancer Sci. 2013 Apr;104(4):465-72. doi: 10.1111/cas.12106. Epub 2013 Mar 7. PMID 23331518
- [Derived] Murata S, Shirakawa M, Sugawara Y, Shuto M, Sawata M, Tanaka Y. Post-hoc analysis of injection-site reactions following vaccination with quadrivalent human papillomavirus vaccine in Japanese female clinical trial participants. Papillomavirus Res. 2020 Dec;10:100205. doi: 10.1016/j.pvr.2020.100205. Epub 2020 Aug 19. PMID 32827835

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 14 sites in Japan from 2006 to 2009.
Pre-assignment Details: There were no specific criteria.
Groups:
- V501: V501; Gardasil, 0.5 mL intramuscular injection, in 3 dosing regimen, given at Day 1, Month 2, and Month 6
- Placebo: Placebo 0.5 mL intramuscular injection, in 3 dosing regimen, given at Day 1, Month 2, and Month 6
Period: Overall Study
Arm/Group | V501 | Placebo
Started | 509 | 512
Vaccinated | 509 | 512
Completed | 453 | 454
Not Completed | 56 | 58
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 24 | 29
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 17 | 21
Not completed — Moved | 4 | 3
Not completed — Pregnancy | 7 | 5
Not completed — Laboratory test values abnormal | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | V501 | Placebo | Total
Number analyzed (Participants) | 509 | 512 | 1021
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.7 (2.1) | 22.9 (2.1) | 22.8 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 509 | 512 | 1021
  Male | 0 | 0 | 0
Body Weight [Mean (Standard Deviation); unit: Kilograms] | 52.1 (8.2) | 51.7 (7.3) | 51.9 (7.8)

OUTCOME MEASURES:

1. Primary Outcome: Combined Incidence of Persistent Human Papillomavirus (HPV) 6, 11, 16 and 18 Infection or HPV 6, 11, 16 and 18 Related-Disease as Determined by Clinical/Pathologic Criteria and Positive Polymerase Chain Reaction (PCR) Assay for Virus Subtype
Description: Participants with HPV 6, 11, 16 or 18 persistent infection, and genital disease (e.g., cervical, vaginal or vulval intraepithelial neoplasia, or cancer, adenocarcinoma in situ and genital warts) per 100 person-years of follow up.
Time Frame: Over 30 months
Population: Includes participants who were not general protocol violators, received all 3 vaccinations, and were seronegative at Day 1 and PCR negative through Month 7 for the relevant HPV type
Measure: Number; unit: Incidence per 100 person-years
Arm/Group | V501 | Placebo
Number analyzed (Participants) | 419 | 422
Incidence per 100 person-years | 0.4 [61.2 to 97.7] | 3.1 [0.0 to 0.0]
Statistical Analysis 1: Comparison: V501 vs Placebo; Test type: Superiority or Other; Percent Relative Risk Reduction = 87.6, 95% CI 2-sided [59.2 to 97.6] — Binomial probability conditional on the fixed number of events

2. Secondary Outcome: Vaccine Type Serum Antibody Titer at One Month After Completed Vaccination Series (Anti-HPV 6)
Description: Month 7 HPV Competitive Luminex immunoassay (cLIA) Geometric Mean Titers (GMTs) by vaccine group.
  The limit of detection of the assay was 7 mMU/ml. GMTs and confidence limits below the limit of detection are shown as "7.0".
Time Frame: At one month after completed vaccination series (Month 7)
Population: Includes participants who were not general protocol violators, received all 3 vaccinations within acceptable day ranges, were seronegative at Day 1 for the relevant HPV type, and had a Month 7 serum sample collected within an acceptable time range
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Titers
Arm/Group | V501 | Placebo
Number analyzed (Participants) | 386 | 365
Geometric Mean Titers | 390.8 [357.7 to 426.9] | 7.0 [7.0 to 7.0]
Statistical Analysis 1: Comparison: V501 vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Vaccine Type Serum Antibody Titer at One Month After Completed Vaccination Series (Anti-HPV 11)
Description: Month 7 HPV cLIA Geometric Mean Titers by vaccine group.
  The limit of detection of the assay was 8 mMU/ml. GMTs and confidence limits below the limit of detection are shown as "8.0".
Time Frame: At one month after completed vaccination series (Month 7)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Titers
Arm/Group | V501 | Placebo
Number analyzed (Participants) | 386 | 365
Geometric Mean Titers | 579.8 [538.1 to 624.8] | 8.0 [8.0 to 8.0]
Statistical Analysis 1: Comparison: V501 vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Vaccine Type Serum Antibody Titer at One Month After Completed Vaccination Series (Anti-HPV 16)
Description: Month 7 HPV cLIA Geometric Mean Titers by vaccine group.
  The limit of detection of the assay was 11 mMU/ml. GMTs and confidence limits below the limit of detection are shown as "11.0".
Time Frame: At one month after completed vaccination series (Month 7)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Titers
Arm/Group | V501 | Placebo
Number analyzed (Participants) | 357 | 365
Geometric Mean Titers | 2396.4 [2201.3 to 2608.8] | 11.0 [11.0 to 11.0]
Statistical Analysis 1: Comparison: V501 vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Vaccine Type Serum Antibody Titer at One Month After Completed Vaccination Series (Anti-HPV 18)
Description: Month 7 HPV cLIA Geometric Mean Titers by vaccine group.
  The limit of detection of the assay was 10 mMU/ml. GMTs and confidence limits below the limit of detection are shown as "10.0".
Time Frame: At one month after completed vaccination series (Month 7)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Titers
Arm/Group | V501 | Placebo
Number analyzed (Participants) | 389 | 386
Geometric Mean Titers | 369.0 [335.9 to 405.4] | 10.0 [10.0 to 10.0]
Statistical Analysis 1: Comparison: V501 vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Serious adverse event data were collected over the entire duration of the study. Other non-serious adverse event data were collected from Day 1 to Day 15 following vaccination.
Description: The number of subjects at risk included randomized participants who had follow-up after at least one dose of vaccine.
  Unlike many countries, in Japan high-grade cervical intraepithelial neoplasias (eg, cervical dysplasia) are often treated in the hospital and are thus categorized as serious adverse events.
Arm/Group | V501 | Placebo
Serious Adverse Events (participants affected / at risk) | 39/480 | 65/468
Other Adverse Events (participants affected / at risk) | 435/480 | 396/468
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V501 (N=480) | Placebo (N=468)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hernia (General disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Meningitis aseptic (Infections and infestations) | 1 (1) | 0 (0)
Ovarian abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Drug toxicity (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Neck injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 1 (2)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 20 (20) | 46 (46)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Abortion induced (Surgical and medical procedures) | 1 (1) | 3 (3)
Ovarian cystectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Tonsillectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1)
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V501 (N=480) | Placebo (N=468)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Palpitations (Cardiac disorders) | 0 (0) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Asthenopia (Eye disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 2 (2)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 1 (1) | 1 (1)
Keratitis (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 3 (3)
Abdominal pain lower (Gastrointestinal disorders) | 3 (3) | 5 (5)
Abdominal pain upper (Gastrointestinal disorders) | 9 (12) | 8 (11)
Constipation (Gastrointestinal disorders) | 0 (0) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 12 (12) | 9 (10)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hyperchlorhydria (Gastrointestinal disorders) | 2 (2) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 11 (11) | 13 (15)
Stomach discomfort (Gastrointestinal disorders) | 6 (6) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 6 (6) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3)
Chest pain (General disorders) | 1 (1) | 1 (1)
Face oedema (General disorders) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 1 (1)
Injection site anaesthesia (General disorders) | 2 (3) | 3 (3)
Injection site bruising (General disorders) | 1 (1) | 3 (3)
Injection site discolouration (General disorders) | 1 (1) | 0 (0)
Injection site discomfort (General disorders) | 8 (12) | 3 (3)
Injection site erythema (General disorders) | 147 (206) | 99 (154)
Injection site haemorrhage (General disorders) | 15 (16) | 1 (1)
Injection site induration (General disorders) | 2 (2) | 1 (1)
Injection site movement impairment (General disorders) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 397 (867) | 316 (626)
Injection site paraesthesia (General disorders) | 0 (0) | 2 (2)
Injection site pruritus (General disorders) | 25 (29) | 11 (12)
Injection site rash (General disorders) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 2 (2)
Injection site swelling (General disorders) | 123 (188) | 57 (84)
Injection site warmth (General disorders) | 3 (4) | 3 (3)
Malaise (General disorders) | 14 (16) | 16 (18)
Puncture site pain (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 39 (40) | 28 (29)
Swelling (General disorders) | 1 (1) | 1 (1)
Venipuncture site swelling (General disorders) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 2 (2) | 7 (7)
Dental caries (Infections and infestations) | 2 (2) | 2 (2)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Laryngopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Lymph gland infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 52 (59) | 52 (60)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (3) | 0 (0)
Purulence (Infections and infestations) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 1 (2)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 3 (3)
Vaginal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 2 (2) | 3 (5)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury corneal (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (3) | 6 (6)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 2 (2)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (2)
Blood pressure decreased (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Glucose urine present (Investigations) | 1 (1) | 2 (2)
Haematocrit decreased (Investigations) | 1 (1) | 3 (3)
Haemoglobin decreased (Investigations) | 0 (0) | 4 (4)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Platelet count increased (Investigations) | 0 (0) | 3 (3)
Protein total decreased (Investigations) | 0 (0) | 2 (2)
Protein urine present (Investigations) | 2 (2) | 6 (6)
Red blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 3 (3)
Weight increased (Investigations) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 1 (1)
White blood cell count increased (Investigations) | 4 (4) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 5 (5) | 6 (8)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 62 (74) | 50 (67)
Hyperaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 3 (3)
Migraine (Nervous system disorders) | 0 (0) | 2 (2)
Somnolence (Nervous system disorders) | 2 (2) | 3 (4)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 1 (1)
Dysphoria (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1)
Neurogenic bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Cervix haemorrhage uterine (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 16 (17) | 28 (34)
Genital pruritus female (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 2 (2) | 4 (4)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (6)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Comedone (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Eczema (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (5)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Urticaria generalised (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.